CLINICAL TRIAL: NCT02850614
Title: Incentivizing Physical Activity Using Gamification, A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: GameTheory (Unknown)
Responsible Party: Principal Investigator, Lizzy Pope, Assistant Professor and DPD Director, University of Vermont
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-080
Record Dates: First submitted 2016-07-26; First posted 2016-08-01 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Physical Activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Fifty participants in the control condition will each receive a FitBit to track their physical activity. Instead of interfacing with a gaming app on their Chromebooks to track physical activity, control condition participants will interface with a minimalist activity tracker showing them only how many minutes of MVPA they've done over the course of the day. It is expected that after several weeks of baseline use, control condition participants will no longer find the FitBit novel. In order to encourage control condition participants to wear their FitBits at school daily, they will receive one entry into a weekly lottery for each day they wear the FitBit that week.
  Interventions: Device: FitBit
- Intervention (Experimental): Fifty participants will be randomized to the intervention condition, which will use a gaming application to encourage physical activity, as physical activity goal achievement will translate into rewards in the game. Physical activity will be tracked using a FitBit activity monitor and in order to encourage intervention condition participants to wear their FitBits at school daily, they will receive one entry into a weekly lottery for each day they wear the FitBit that week.
  Interventions: Behavioral: gaming application to encourage physical activity; Device: FitBit

INTERVENTIONS:
Behavioral: gaming application to encourage physical activity
  Arms: Intervention
Device: FitBit

SUMMARY:
Juniors and seniors will be recruited to participate in the study, which will begin in the fall 2016 and run through May. The intervention will be a randomized-controlled trial, where students are randomized to either a control or incentive condition. Physical activity will be automatically tracked throughout the study period using FitBit activity trackers wirelessly linked to the gaming application on students' Chromebooks or mobile phones. Students who achieve 30 minutes of MVPA during the school day and/or 60 minutes of MVPA over the entire day will receive in-game rewards moving them up leaderboards in the game, providing them with more game points, or allowing them access to more game elements. Baseline outcome measures will be collected at the beginning of the school year in the fall, and post-intervention outcome measures will be collected in May.

DETAILED DESCRIPTION:
Physical Activity Goals and Options Two physical activity goals will be reinforced during the intervention. First, reinforcement will be delivered contingent on achieving the CDC target of 60 minutes of moderate and vigorous physical activity (MVPA) over the whole day. Because in-school activity is important for student health, participants will also earn in-game reinforcement for achieving 30 minutes of MVPA during the school day as targeted by the VT State Board of Education. Students who meet both goals will receive the most in-game rewards.

In order to help students achieve the physical activity targets, opportunities for completing short bouts of physical activity or taking extra steps throughout the school day and before/after school will need to be offered. Youth input as well as BHS teacher and staff input will be integral in determining which types of additional activity opportunities are feasible. Other Vermont schools have integrated physical activity into Teacher Advisor time as well as offering physical activity breaks during or between academic classes. Active transport to school, or taking advantage of before and after school activity options already offered at BHS will be additional ways for students to meet the 60 minutes/day target. The gamification aspect of the intervention will allow students to use the layout of BHS to accumulate more minutes of physical activity throughout the day. Students will be able to check-in at various locations around the high school using QR codes to earn physical activity points in the game. MVPA accumulation will be tracked automatically using a FitBit, which indicates the number of minutes the student was active at a moderate or vigorous level during the day. The FitBit will then automatically and wirelessly communicate with the gaming app on the student's Chromebook to determine the quantity of game rewards awarded daily. Rewards will be available immediately upon meeting MVPA goals.

Mobile Game Incentivizing Physical Activity The specific elements to be used in the game have been determined by conducting focus groups with BHS sophomores and juniors as well as working with the game developers, GameTheory, a local game development company with experience designing games that transform tedious tasks into fun ones (gametheoryco.com). Basic game theory suggests certain gaming elements that are especially effective at encouraging engagement, which will be incorporated into the game design. Elements of effective games such as self-representation with avatars, 3D environments, narrative context, unpredictability, leaderboards, options to work in teams or clans, and check-in based mechanisms where the game continues to evolve even when the player is not logged in are all aspects of our game design. Furthermore, the game design incorporates theories of behavioral economics that can be capitalized on in a game environment such as present-bias and loss aversion. Lastly, principles of monetary incentive interventions successfully used to promote sustained accomplishment of various health behaviors in previous research, such as escalating rewards with a reset contingency for missed goals and random ratio reinforcement schedules are integrated. Game "points" will be awarded for achieving the two physical activity daily goals, with an extra daily bonus for meeting both goals.

The premise of the game is that students are involved in a water balloon clash at a woodsy-feeling summer camp. Each week, participants will be divided into two "teams" who will engage in a series of water balloon clashes during the week. Students will be able to customize an avatar that represents them during the game. They will be able to select an avatar name (which will be approved by investigators before becoming active), as well as customize the look of their character. Furthermore, they will be able to see their character's "stats" in terms of how strong, how healthy, and how much speed their character has. The amount of physical activity participants record on their FitBit each day will determine how much their character's stats improve from day to day. Students will be rewarded for recording real-world physical activity on their FitBits with the translation of steps they take into "coins" which students can use to buy items for their avatars. Items coins can purchase will include supplies for upcoming water balloon clashes, costumes and special clothing pieces like sneakers, healthy snacks, and pets. Therefore, students will be able to create a customized world for their characters using the coins they earn from their real-world steps. Students will also be rewarded for improvements in their physical activity status, being top physical activity performers, and meeting the two daily physical activity goals in the form of gems. On certain days, multiple gems will be given for meeting goals, providing a random bonus that will serve as variable-interval reinforcement for game players. Therefore, every step participants take with their FitBit lets them obtain coins in the game, whereas meeting the bigger goals or showing improvement will earn participants gems, which have a higher value than coins.

Each day, the game will automatically run a water balloon skirmish between the two teams' treehouses. Students will choose where to position their avatar for attack or defense, and see where their teammates are positioned. The game will then use an algorithm based on the avatars' positions as well as the accumulated strength, speed, and health of the various avatars on each team to determine which team wins the daily battle. Students can then log-in and watch replays of the battle as well as see the results in terms of which team got hit the most, how many water balloons their avatar threw, how many defensive actions they successfully carried out, and who on the other team hit them with a water balloon. Students will receive in-game prizes or gems for achieving certain milestones throughout the clash such as being the "Best defender," "Most balloons landed," etc. Teams will aim to win the most clashes each week, and then the teams will be reshuffled.

ELIGIBILITY:
Inclusion Criteria:

* 15-18 years of age Junior or Senior at Target High School BMI >=18.5

Exclusion Criteria:

* Current participation in a formal weight-loss program Physical activity limitations

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Physical Activity - Steps | 12 weeks
  The primary measurement tool for physical activity will be the use of FitBits to quantify the number of minutes students are moving each day, and the number of steps they are taking. Even the most basic FitBits capture steps, distance, minutes people are active each day, and intensity of activity. They are then able to wirelessly sync with the study database and gaming application (intervention condition) or tracking application (control condition), so accounting for activity will be automatic. FitBits have been validated as an acceptable measurement tool for measuring physical activity in free-living individuals.48 It is anticipated that most physical activity students engage in would be traceable with the FitBit. Physical activity in both the control and intervention conditions will be continuously tracked throughout the baseline, intervention, and post-intervention periods.
Physical Activity - Minutes of Moderate or Vigorous Physical Activity | 12 weeks

SECONDARY OUTCOMES:
Height | Baseline and at 12 weeks
Student Engagement | Baseline and at 12 weeks
  Student engagement will be assessed at baseline and post-intervention using a self-administered previously established student engagement scale assessing student connectedness and whole-school connectedness. The scale was developed by Bradshaw et al., as part of the Maryland Safe and Supportive School Climate Survey.49 This scale includes 9-items with 4-point Likert scale response options.
Weight | Baseline and at 12 weeks
BMI | Baseline and at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will deposited in a repository after the study is finished.